CLINICAL TRIAL: NCT00235586
Title: Vitamin D Deficiency: Bone Loss and Vascular Dysfunction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Kansas (Other)
Collaborators: National Osteoporosis Foundation (Other)
Organization: University of Kansas Medical Center (Other)
Allocation: Non-Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: 9248
Record Dates: First submitted 2005-10-06; First posted 2005-10-10 (Estimated); Last update posted 2007-09-20 (Estimated); Status verified 2007-09

CONDITIONS: Postmenopausal Women
Keywords: vitamin D deficiency postmenopausal women

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: 10 vit. D deficient subjects take vit. D for 3 months.

SUMMARY:
To learn if there is a connection between low vitamin D level and hardening of the arteries.

DETAILED DESCRIPTION:
Osteoporosis and vascular disease are two of the most common disorders affecting postmenopausal women. A potential association, beyond aging, has long been speculated. Our previous study revealed evidence of loss of vascular compliance in postmenopausal women with lower bone density, suggesting women with lower bone density had "stiffer" blood vessels. This proposal further investigates that association and a potential role of vitamin D deficiency as a possible common link between both bone loss and "hardening of the arteries".

ELIGIBILITY:
Inclusion Criteria:

* Females ages 50-70 with ability to give informed consent
* One year past last menstrual period
* 20 women with Vitamin D levels < 15 mg/ml
* 20 women with Vitamin D levels > 30 mg/ml

Exclusion Criteria:

* women receiving hormone replacement therapy
* women receiving medication known to effect vascular compliance, including anti-hypertension medications
* subjects receiving therapy for osteoporosis
* hyperthyroidism
* untreated hypothyroidism
* history of metabolic bone disease
* current or previous use of medications known to accelerate bone loss
* chronic liver disease
* chronic renal disease
* diabetes mellitus
* obesity, BMI > 24

Ages: 50 Years to 90 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40
Dates: Start 2004-04; Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
to determine if differences exist in vascular compliance and carotid artery intima media thickness between individuals with normal and low vitamin D levels
to evaluate correlation of markers of vascular disease and boen disease between individuals with normal and low vitamin D
to quantify the effect of Vitamin D replacement on vascular compliance and markers of bone loss and vascular disease.

SECONDARY OUTCOMES:
Vitamin D at the end of 3 months of supplementation.

CONTACTS AND LOCATIONS:
Overall Officials: Leland Graves, III, MD, Principal Investigator — University of Kansas Medical Center
Locations (1):
- University of Kansas Medical Center, Kansas City, Kansas, United States